CLINICAL TRIAL: NCT06566326
Title: Oropharyngeoesophageal Topical Anesthesia Prototype Device Versus Intravenous (Propofol - Ketamine Sedation) for Upper Gastrointestinal Endoscopy
Brief Title: Oropharyngeoesophageal Topical Anesthesia Versus Propofol - Ketamine Sedation for Upper Gastrointestinal Endoscopy
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Zagazig University (Other Government)
Responsible Party: Principal Investigator, Ashraf Torki, Lecturer of Anesthesia, Zagazig University, Zagazig University
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: ZU-IRB #10002
Record Dates: First submitted 2024-08-20; First posted 2024-08-22 (Actual); Last update posted 2024-08-30 (Actual); Status verified 2023-07

CONDITIONS: Upper Gastrointestinal Endoscopy; Topical Anesthesia; Intravenous Sedation
Keywords: Topical Anesthesia; Upper Gastrointestinal Endoscopy; Propofol - ketamine sedation
MeSH Terms: interventions — Propofol; Ketamine

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Group (PK) (Active Comparator): Patients received intravenous sedation using prepared mixture of propofol and ketamine (in the ratio 4:1)
  Interventions: Drug: Propofol and ketamine
- Group (OPETA) (Active Comparator): Patients underwent modified Oropharyngeo-esophygeal Topical Anesthesia by OPETA Prototype tool
  Interventions: Device: Modified Oropharyngeo-esophygeal Topical Anesthesia by OPETA Prototype tool

INTERVENTIONS:
Drug: Propofol and ketamine — Patients received IV sedation using prepared mixture of propofol and ketamine in ratio (4:1). It is prepared by mixing 0.8 mg/kg propofol with 0.2 mg/kg ketamine (4:1) in an IV bolus, followed by half of the initial dose every 3 minutes as needed for sedation. The desired level of sedation was achieved (more than score 4) using Modified Ramsay sedation score) before allowing endoscopiest to start the procedure, then the score was assessed every 3 minutes before giving of top up doses of ketofol 4:1 (half of the initial dose) if needed, then the range and median of modified Ramsay sedation score was calculated.
  Other Names: Intravenous sedation
  Arms: Group (PK)
Device: Modified Oropharyngeo-esophygeal Topical Anesthesia by OPETA Prototype tool — Topicalization was done for anterior tonsillar pillar on both sides and posterior 1/3 of tongue and posterior pharyngeal wall using xylocain gel 5 % on tip of his index or middle finger then after 5-7 min. patient inserted his middle finger deeply into his mouth as a test for tolerability before insertion of OPETA tool. While head tilted forward, Lubricated OPETA device, soaked with 10 ml lidocaine 2 % mixed with adrenaline 1/200000 was gradually placed by patient with assistance from anesthetist & patients swallowing into esophagus. To ensure effective topical anesthesia and patient tolerance, pack was left in place for 3-5 min. before being moved up, down, clockwise & anti-clockwise.. If necessary, increments of 5 ml of 2% lidocaine/adrenaline mixture was injected through device until patient is comfortable. Maximum LA dose was kept at 5 mg/kg.
  Arms: Group (OPETA)

SUMMARY:
Esophagogastroduodenoscopy (EGD) is an essential and widely used diagnostic and therapeutic procedure in gastroenterology. EGD can be performed in association with topical anesthesia of the pharynx, intravenous anesthesia, or with their combination. Sedation is required to alleviate anxiety, provide analgesia, amnesia and to improve endoscopic performance specifically in therapeutic procedures. However, sedation-related gastrointestinal endoscopy complications when occur, may lead to significant morbidity and occasional mortality especially with moderate and deep sedation. Cardiopulmonary complications resulting from aspiration, oversedation, hypoventilation, vasovagal reflex, and airway obstruction account for more than 50% of all complications associated with upper endoscopy. Topical pharyngeal anesthesia currently is a requirement for upper endoscopy to provide patients with the best comfort in unsedated EGD. In Hong Kong, 10% Xylocaine pump spray (AstraZeneca, Sodertalje, Sweden) is the pharyngeal anesthesia generally used as a premedication in unsedated EGD. The aim of this study was to provide more effective, safer, tolerable and offers quicker recovery technique using either the modified Oropharyngeoesophageal Topical Anesthesia (OPETA) technique or conventional intravenous sedation by prepared mixture of propofol and ketamine (ketofol 4:1) .

DETAILED DESCRIPTION:
This Randomized prospective clinical study was conducted at Zagazig University Hospitals in anesthesia, intensive care and pain management department at the outpatient endoscopy unit service at general medicine department on 60 patients scheduled to undergo elective upper GI endoscopy. All upper GI endoscopy procedures was preformed by OLYMPUS EVIS EXERA III CV- 190 .Written informed consent was obtained from all participants.

According to a computer-generated randomization table, patients were allocated to two equal groups (30 patients in each group). Group (PK): Included 30 patients received intravenous sedation using prepared mixture of propofol and ketamine (in the ratio 4:1).

Group (OPETA):

Included 30 patients underwent modified Oropharyngeo-esophygeal Topical Anesthesia by OPETA Prototype tool (Nofal 2010).

All participants were subjected to:

Obtaining of history and physical examination including vital signs, cardiac and chest condition as well as excluding criteria. Routine laboratory investigations included Complete blood count (CBC), Random blood sugar, coagulation profile (PT, PTT, INR) liver function tests , renal function tests . General and airway examination was done All patients were kept fasting for 4 hours from clear fluids and 6 hours from other foods Midazolam 2-2.5 mg IV was given to all patients at holding area.

Study design:

After routine pre-operative evaluation, standard monitors were connected to the patients: pulse oximetry, noninvasive blood pressure and electrocardiogram and baseline parameter were recorded (peripheral oxygen saturation, mean arterial pressure and heart rate). Intravenous (IV) line will be inserted and atropine IV 1 mg administered for all patients. Patients will be allocated into two equal groups by a computer-generated randomization table:

Group (PK) (n=30):

Patients received intravenous sedation using prepared mixture of propofol and ketamine in ratio (4:1). It is prepared by mixing 0.8 mg/kg propofol with 0.2 mg/kg ketamine (4:1) in an IV bolus, followed by half of the initial dose every 3 minutes as needed for sedation. The desired level of sedation was achieved (more than score 4) using Modified Ramsay sedation score) before allowing endoscopiest to start the procedure, then the score was assessed every 3 minutes before giving of top up doses of ketofol 4:1 (half of the initial dose) if needed, then the range and median of modified Ramsay sedation score was calculated.

Group (OPETA) (n=30):

Every patient by him or herself or by help of anesthetist topicalized the anterior tonsillar pillar on both sides and the posterior one third of the tongue as well as the posterior pharyngeal wall using xylocain gel 5 % on the tip of his index or middle finger then after 5-7 minutes the patient inserted his middle finger deeply into his mouth as a test for tolerability before the insertion of OPETA tool (the patient was instructed not to swallow the used local anesthetic but gurgle it as long as possible). While the head tilted forward ("chin on chest"), Lubricated Oropharyngeoseogageal pack (OPETA device), soaked with 10 ml lidocaine 2 % mixed with adrenaline 1/200000 was gradually placed by the patient himself or herself with assistance from the anesthetist and patients swallowing into the esophagus. To ensure effective topical anesthesia and patient tolerance, the pack was left in place for three to five minutes before being moved up, down, clockwise and anti-clockwise.. If necessary, increments of 5 ml of 2% lidocaine/adrenaline mixture was injected through the device until the patient is comfortable. For all patients, the maximum local anesthetic dose (5 mg/kg of lidocaine without adrenaline and 7 mg/kg of a lidocaine with adrenaline 1:200000) was meticulously considered. However, we tryied to keep the maximum dosage at 5 mg/kg as we dealing with topical anesthesia at the mucous membrane.

The Oropharyngeo-esophygeal Topical Anesthesa (OPETA) device:

It is a handmade device of a patented concept (patency no 23733, academy of scientific research and technology, ARST. Egypt, it is originally used as supraglottic topical anesthesia device. The prototype OPETA device consists of orogastric tube surrounded by a cotton gauze of 5 cm. width. The tube and device size are age dependent and usually of 16-gauge tube size. The tip of the orogastric tube is burnt e.g., by a flame of lighter and simultaneously clamped by a needle holder. Air under pressure is then pushed through the tube port using a 10 ml syringe to verify integrity of the closed tip. Starting from the burnt closed tip, the orogastric tube was punctured with a 21-gauge needle in two perpendicular planes with 1 cm in between each puncture within the same plane for 45 to 50 cm in adult cases representing the length of a line passing from the mouth to earlobe then to xyphoid process. 5 cm wide cotton gauze was wrapped over the punctured part of the tube and secured with 2- 0 Mersilk. After inserting the device into the oropharyngeal cavity and esophagus, local anesthetic (LA) /adrenaline mixture was injected into the punctured tube when required. The injected LA was sprayed through the puncture sites to the surrounding cotton gauze that is in contact with the oropharyngeal and esophageal mucosa, anesthetizing it. During the device insertion, if it is required to make the device less malleable for easier insertion, part of an ureteric guide wire or ureteric catheter cover could be inserted within the tube of the device to strengthen it. After getting the patient sedated or topically anesthetized, endoscopist started the procedure. The modified Aldrete's scoring system was used for the discharge of all patients from recovery. Achievement of at least 9 out of 10 scores was the criteria for discharge in this study. Twenty four hour after the procedure all patients were asked through telephone connection about their experiences regarding the intraprocedural events, they were asked to score their satisfaction level during the procedure in terms of recalling any painful or other undesirable intraprocedural events.

Monitoring:

Standard monitors for all cases include patient's heart rate, oxygen saturation, and MAP pre-procedural (basal) for both topical and sedation groups then every 5 minutes throughout the procedure until the patient is fully alert. Side effects such as hypotension and bradycardia were recorded, if hypotension occurs (decrease in MAP more than 20% from baseline) it was treated with normal saline and if blood pressure was not corrected, ephedrine 5 mg was administered incrementally, and if bradycardia occurs (HR < 60 beats/min) it was treated with atropine 0.01 mg/kg).

Post procedural assessment:

1. Patient assessment:

   * Two separate questionnaires were asked to the patients in order to rate the procedure 24 hours after discharge when they become completely alert (through telephone connection). The patients answered the following questions:
   * The difficulty in insertion of OPETA device.
   * Discomfort they felt during procedure. Answers was given on a 0 -10-mm numeric rating scale. The left end of the scale (0 mm) will be defined as ''not at all'' and the right end (10 mm) as ''extremely.
2. Endoscopist assessment:

The endoscopist assessed the following:

1. Difficulty in introducing the endoscope.
2. The overall technical difficulty of the examination.
3. Gagging whether occurred or not. For endoscopist's assessment the 0-10 numeric rating scale was the measurement scale where 0 means the procedure was extremely comfortable and 10 means that it was extremely uncomfortable.

Data collection:

Patient characteristics (Age, Sex, ASA physical status class, BMI). Indications of endoscopic procedure. Baseline heart rate, mean arterial blood pressure (MAP), and oxygen saturation were recorded every five minutes throughout endoscopic procedure and every 10 minutes when the patients at PACU. Patient Assessment: numeric rating scale (0 …………..…….10)

1. Discomfort felt during the procedure.
2. Willing to Re-do in OPETA group. Endoscopist Assessment: numeric rating scale (0 …………….. 10) 1. Difficulty in introducing the endoscope. 2. Gagging with esophageal intubation. 3. The endoscopist satisfaction. Number of doses in PK group.

Time:

1. OPETA time: Time from administration of self or helped oral topical anesthesia till getting the OPETA device manipulation tolerated by the patient (moving the OPETA tool up and down clockwise and anti-clockwise without distressing the patient).
2. Sedation time: Time from starting intravenous sedation until ability to insert endoscope freely.
3. Endoscopy time: Time from starting of insertion till removal of the endoscope.
4. Recovery time: Time since the endoscopist finish the endoscopy until the patient is completely alert and oriented to space and time.
5. Discharge time: Time from admission to the recovery area to get the patient ready for discharge from the recovery area using modified aldert score.
6. Total time: summation of previous times. Any complications e.g., systemic toxicity, respiratory depression, desaturation, nausea and vomiting in both studied groups were recorded and managed.

ELIGIBILITY:
Inclusion Criteria:

Both sexes. Patients aged between 21-64 years old undergoing elective upper GI endoscopy after taking informed consent. ASA class II /III BMI < 30kg/m2

Exclusion Criteria:

Hypersensitivity to drugs included in the study. Difficult airway or known airway problems. Active bleeding from esophageal varices. Emergency procedure Low base line oxygen saturation < 92% at room air. Cases expected to need general anesthesia for the procedure as judged by endoscopist.

Ages: 21 Years to 64 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 60 (Actual)
Dates: Start 2023-01-01 (Actual); Primary Completion 2023-07-01 (Actual); Study Completion 2023-07-30 (Actual)

PRIMARY OUTCOMES:
Patient discomfort felt during endoscopy | Endoscopy time: Time from starting of insertion till removal of the endoscope
  0-10 numeric rating scale was the measurement scale where 0 means the procedure was extremely comfortable and 10 means that it was extremely uncomfortable.

SECONDARY OUTCOMES:
Difficulty in insertion of OPETA device | OPETA time: Time from administration of self or helped oral topical anesthesia till getting the OPETA device manipulation tolerated by the patient (moving the OPETA tool up and down clockwise and anti-clockwise without distressing the patient).
  0-10 numeric rating scale was the measurement scale where 0 means the procedure was extremely comfortable and 10 means that it was extremely uncomfortable.
Difficulty in introducing the endoscope | Endoscopy time: Time from starting of insertion till removal of the endoscope
  0-10 numeric rating scale was the measurement scale where 0 means the procedure was extremely comfortable and 10 means that it was extremely uncomfortable.
Overall technical difficulty of the examination | Endoscopy time: Time from starting of insertion till removal of the endoscope
  0-10 numeric rating scale was the measurement scale where 0 means the procedure was extremely comfortable and 10 means that it was extremely uncomfortable.

CONTACTS AND LOCATIONS:
Overall Officials: Osama A Nofal, MD, Study Director — Zagazig University; Rania A Kamel, MD, Study Chair — Zagazig University; Badiea B Elhag, Msc, Principal Investigator — Zagazig University
Locations (1):
- Zagazig university hospitals, Zagazig, Sharqia Province, Egypt

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Amornyotin, S. (2015). Anesthesia innovations for endoscopy of gastrointestinal tract. Endoscopy-innovative uses and emerging technologies. Croatia: InTech, 39-61.
- [Background] de la Morena F, Santander C, Esteban C, de Cuenca B, Garcia JA, Sanchez J, Moreno R. Usefulness of applying lidocaine in esophagogastroduodenoscopy performed under sedation with propofol. World J Gastrointest Endosc. 2013 May 16;5(5):231-9. doi: 10.4253/wjge.v5.i5.231. PMID 23678376
- [Background] hfeda, M. A. M., Ganaw, A., Ahmed, S. M. G., Chanda, A., Mahood, Z., Jabira, S., et al . (2021). Anaesthetic Considerations in Gastrointestinal Endoscopies. In Esophagitis and Gastritis-Recent Updates. (Edited by Vincenzo Neri and Monjur Ahmed) Ch 9, P. 141- 158. BoD- Book on Demand .
- [Background] Feng AY, Kaye AD, Kaye RJ, Belani K, Urman RD. Novel propofol derivatives and implications for anesthesia practice. J Anaesthesiol Clin Pharmacol. 2017 Jan-Mar;33(1):9-15. doi: 10.4103/0970-9185.202205. PMID 28413268
- [Background] Heuss LT, Hanhart A, Dell-Kuster S, Zdrnja K, Ortmann M, Beglinger C, Bucher HC, Degen L. Propofol sedation alone or in combination with pharyngeal lidocaine anesthesia for routine upper GI endoscopy: a randomized, double-blind, placebo-controlled, non-inferiority trial. Gastrointest Endosc. 2011 Dec;74(6):1207-14. doi: 10.1016/j.gie.2011.07.072. Epub 2011 Oct 13. PMID 22000794
- [Background] Kamalipour, H., Joghataei, P., & Kamali, K. (2009). Comparing the Combination Effect of Propofol-Ketamine and Propofol-Alfentanil on Hemodynamic Stability during Induction of General Anesthesia in the Elderly.
- [Background] Nofal O. Awake light-aided blind nasal intubation: prototype device. Br J Anaesth. 2010 Feb;104(2):254-9. doi: 10.1093/bja/aep367. Epub 2009 Dec 26. PMID 20037149